CLINICAL TRIAL: NCT04815135
Title: The Impact Of The Covid-19 Pandamic On Emergency Surgery In A Tertiary Hospital In Jordan. A Cross Sectional Study
Brief Title: Effect of Covid-19 Pandemic on Emergency Surgery Practice
Status: Completed | Type: Observational
Sponsor: Ibrahim Khrais (Other)
Responsible Party: Sponsor-Investigator, Ibrahim Khrais, Co-investigator, University of Jordan
Organization: University of Jordan (Other)
Other Study IDs: 10-2021-5926
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Emergencies
MeSH Terms: conditions — Emergencies | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 2020 group (COVID19 group): Patients who were admitted to the surgical ward via the emergency department during the lockdown period due to the COVID19 pandemic
  Interventions: Other: Observational study
- 2019 group (pre COVID19 group): Patients who were admitted to the surgical ward via the emergency department during the similar period in 2019

INTERVENTIONS:
Other: Observational study — Observational study, the study did not involve any interventions
  Groups: 2020 group (COVID19 group)

SUMMARY:
A retrospective study at a tertiary university hospital to determine the effect of the COVID-19 pandemic on the emergency surgery practice in the hospital.

DETAILED DESCRIPTION:
The investigators conducted a retrospective review of all the patients who were admitted to the surgical wards through the emergency department at the Jordan University Hospital in the periods from March 2020 to May 2020. The records were compared to those of the patients who were admitted in the same period from the year 2019.

Data collection includes the number of admissions, the reason for admission, the average of symptoms duration until admission, the age of the patients admitted, gender, type of management, and the average length of stay before discharging the patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients who were admitted to the surgical wards via the emergency department during the study periods

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who were admitted to the surgical wards via the emergency department at our institution.
Sampling Method: Non-Probability Sample
Enrollment: 344 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2021-01-18 (Actual)

PRIMARY OUTCOMES:
Average duration of sx prior to admission in hours | 1 year
Type of management (surgical vs conservative) | 1 year
Length of stays in Days | 1 year
Level of care (ICU vs floor) | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Ibrahim Khrais, Amman, Please Select, Jordan

IPD SHARING:
Plan to Share IPD: Undecided